CLINICAL TRIAL: NCT07327099
Title: Clinical Evaluation of Different Arthrocentesis Techniques in the Treatment of Temporomandibular Joint Disorders
Brief Title: Comparative Assessment of Arthrocentesis Methods in TMJ Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helin Merve Özalp (Other)
Responsible Party: Sponsor-Investigator, Helin Merve Özalp, ressearcher assistant, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTU-DHF-HMO-01
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Joint Disc Displacement, With Reduction
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Arthrocentesis was performed on the first group using a method developed by Mun et al., involving two 22-gauge needles bent to form a 'Y' shape with the tips facing each other, and on the second group using a factory-made Y-shaped cannula developed by Rahal et al.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): The first group underwent arthrocentesis using a method developed by Mun et al., involving two 22-gauge needles bent to form a Y-shape with their angles facing each other.
  Interventions: Procedure: Y-shaped cannula without a source
- group 2 (Active Comparator): The second group underwent arthrocentesis using a method developed by Rahal et al., involving a factory-made Y-shaped cannula.
  Interventions: Procedure: Y-shaped cannula with a source

INTERVENTIONS:
Procedure: Y-shaped cannula without a source — Y-shaped cannula without a source Arthrocentesis performed by simultaneously and concentrically placing two manually Y-shaped bent needles into the joint cavity.
  Arms: group 1
Procedure: Y-shaped cannula with a source — Y-shaped cannula with a source Arthrocentesis performed by simultaneously and concentrically placing two manually Y-shaped bent needles into the joint cavity.
  Arms: group 2

SUMMARY:
Temporomandibular disorders (TMD) are common conditions in society, characterised by symptoms such as pain, limited movement and joint noises, which negatively affect an individual's quality of life. The primary goal of treatment is to restore the physiological functions of the joint by eliminating the aetiological factors. In cases where conservative methods prove ineffective, arthrocentesis, a minimally invasive approach, comes to the fore. Arthrocentesis aims to reduce pain by removing inflammatory mediators and to increase joint mobility. In this study, the intraoperative parameters and clinical outcomes of different arthrocentesis techniques were compared and evaluated in patients with Wilkes stage 2-3 TME disorders.

DETAILED DESCRIPTION:
Introduction: Temporomandibular disorders (TMD) are common symptoms in society, characterized by pain, limited movement, and all sounds, which are often negatively impacted by individual life circumstances. The primary goal of treatment is to eliminate the etiological factors and restore the replaceable functions of the parts. Arthrocentesis, a minimally invasive approach, is emphasized in cases where conservative treatment is beneficial. Arthrocentesis reduces pain by removing inflammatory mediators and increases joint mobility. This effective treatment was evaluated by comparing the intraoperative parameters and clinical success of different arthrocentesis techniques in patients with Wilkes stage 2-3 TMJ disorders.

Materials and Methods: This study is being conducted at the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Karadeniz Technical University. Fifty patients (Group 1: n=25, Group 2: n=25) treated with two different arthrocentesis technologies were enrolled retrospectively. The first group was the study of Mun et al. Arthrocentesis was performed using the method employed by Rahal et al., which consisted of two 22-gauge needles bent to form a "Y" shape and placed simultaneously and concentrically. The second group underwent arthrocentesis using a fabricated Y-shaped cannula used by Rahal et al. Each treatment was performed under local anesthesia, and the upper regions were irrigated with an average of 100 ml of Ringer's lactate solution. Following arthrocentesis, 1 ml of hyaluronic acid was injected into the patients. Preoperative and postoperative values were evaluated by comparing the groups at 1 to 6 months. Furthermore, intraoperative arthrocentesis efficiency (number of needle insertions, procedure time, complication rate, and treatment tolerance) was compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

Patients with unilateral TME disorders who:

* Are in stages 2-3 of the Wilkes classification
* Have not undergone interventional treatment prior to arthroscopy
* Have undergone conservative treatment prior to arthroscopy without successful results

Exclusion Criteria:

* Patients with TME irregularities who have undergone interventional treatment (minimally invasive and invasive)
* Patients with bilateral TME disorders
* Patients with incomplete recorded data

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
TMJ Pain | before the procedure, at 1 month and at 6 months
  Pain was assessed using the VAS scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ktu Dentistry, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared later if required for the confidentiality of the study.

REFERENCES:
- [Result] Senturk MF, Yazici T, Gulsen U. Techniques and modifications for TMJ arthrocentesis: A literature review. Cranio. 2018 Sep;36(5):332-340. doi: 10.1080/08869634.2017.1340226. Epub 2017 Jun 15. PMID 28618972